CLINICAL TRIAL: NCT02129413
Title: Safety and Performance of the Delta System in the Treatment of Vasospasm in Aneurysmal Subarachnoid Hemorrhage (aSAH) Patients
Brief Title: Safety Study of Carotid Body Neurostimulation to Treat Cerebral Vasospasm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samson NeuroSciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLT-CL-PR-01
Record Dates: First submitted 2014-04-24; First posted 2014-05-02 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2014-04

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Cerebral Vasospasm
Keywords: Aneurysmal subarachnoid hemorrhage; Subarachnoid hemorrhage; Cerebral vasospasm; Ruptured aneurysm; Delayed Cerebral Ischemia; Delayed Ischemic Deficit; Delayed ischemic neurological deficit; Neurostimulation; Carotid body
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Aneurysm, Ruptured

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Delta system treatment (Experimental)
  Interventions: Device: Delta system

INTERVENTIONS:
Device: Delta system

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the Delta system in the treatment of cerebral vasospasm post aneurysmal subarachnoid hemorrhage (aSAH) patients.

DETAILED DESCRIPTION:
The Delta system is intended to deliver electrical modulation signal to the carotid body, to result in cerebral vasodilation and blood flow augmentation in the brain, for treatment of patients suffering from vasospasm post aSAH.

In this clinical trial the Delta system in intended to be used on patients who have their ruptured aneurysm secured, hospitalized in the neuro ICU (Intensive Care Unit) and are anesthetized and intubated, diagnose as suffer from cerebral vasospasm, who fulfill all the inclusion criteria and none of the exclusion as detailed in the study protocol.

The system is intended to be used for up to 7 days under hospital supervision that is routinely provided for stabilizing patients following SAH and securing aneurysms. Follow up period is 30 days after end of treatment.

The Delta system is comprised from two main elements: Electrical Stimulation Unit (ESU) and Delivery kit.The ESU is a reusable external autonomic stimulator unit, cable and graphic user interface (GUI) software based on a PC tablet. The delivery kit is a disposable stimulating leads shaft and accessories.

The procedure includes insertion of the leads shaft over a guiding needle via patient neck, so electrodes are positioned adjacent the carotid bodies. Therapy parameters are set by the physician and monitoring is continued during patient hospitalization to determine when therapy can be discontinued and shaft removed.

Twenty three (23) patients will be recruited to the study, including 3 roll-in patients. The study is an open label, uncontrolled, non-randomized, multicenter feasibility study. This study will recruit male and female adult patients with aSAH secondary to rupture of an aneurysm, secured by coiling or clipping, and in WFNS grades I-IV. Only anesthetized and intubated patients will be recruited for the study.

This study evaluates the safety and performance of the Delta system. The potential benefits and risks of participation in this study are clearly identified in the informed consent form and are to be explained to the subject prior to participating in the study.

Study treatment - The Delta system is inserted by minimally exposure of the carotid bifurcation. The system electrically stimulates the carotid body chemoreceptors, aiming to achieve sustainable cerebral vasodilation for inducing enhancement of cerebral perfusion and thereby minimizing ischemia and consequently prevent delayed neurological deficit. Treatment with the delta system is intended for up to seven (7) days.

Manufacturing and assembling the Delta system is done in certified facilities. Further information and complete details regarding device materials, specifications, design, quality assurance, etc. can be found in the Investigator's Brochure.

Risk to benefit rational - reverse vasospasm and increase cerebral blood flow (CBF) is the major component of cerebral perfusion augmentation, results in reducing the rate of vasospasm complication. The Delta system may provide vasospasm subjects with a novel treatment option. Based on the Delta system design, the extensive pre-clinical tests conducted with the system and the comparison to other similar devices and alternative treatments, the company believes that the system is safe for use and beneficial for reduction of delayed cerebral ischemia complication that are vasospasm related.

Statistical analysis plan - Sample size for this study is determined by the secondary end point.

Sample size of N=20 achieves:

* 88% power to detect CBF decrease of ≥ 15% in at least one of the affected cerebral arteries measured by TCD.
* 88% power to detect increase in artery diameter of ≥15% in at least one of the affected main cerebral arteries measured by DSA or CTA.
* 99% power to detect CBF increase of ≥20% measured by CerOx monitor system or Licox® monitoring system.

All with an estimated standard deviation of 0.2 and with alpha of 0.05, using a one-sample t-test analysis. The sample size also serves the qualitative analysis of the primary end point.

A t-test is any statistical hypothesis test in which the test statistic follows a Student's t distribution if the null hypothesis is supported. It can be used to determine if two sets of data are significantly different from each other for continues parameters (such as artery diameter) , and is most commonly applied when the test statistic would follow a normal distribution if the value of a scaling term in the test statistic were known. The estimation for the significant clinical difference as well as the assumed standard deviation was based on previous experience with the device. When the scaling term is unknown and is replaced by an estimate based on the data, the test statistic (under certain conditions) follows a Student's t distribution.

Data management plan - Data management will be directly provided or contracted by the sponsor and compliant to the requirements of ISO 14155:2011. The Sponsor or its designee will provide the investigator with a Case Report Form (CRF) booklet for each subject enrolled in the study and will train the site personnel in the correct manner of recording data. The appropriate CRFs will be completed and signed by the Investigator as appropriate. All CRFs will be completed in a legible manner in blue or black ink. Any corrections will be made by drawing a single line through the incorrect entry, entering the correct information, and initialing and dating the change. Data entry boxes or spaces should not be left blank, but instead should indicate: NA for not applicable, ND for not done or "-"for missing or not available data. The original signed forms, not copies, will be returned to the Sponsor. All clinical data generated in the study will be submitted to the Sponsor or its designee for quality assurance review, data entry, and statistical analysis. All forms will be reviewed for completeness. Any recording errors will be corrected by contact with the appropriate clinical site. Double-entry routines will be utilized to reduce data entry errors, and computerized editing routines will be used to identify unusual data entries for verification prior to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female older than 18 years of age and no more than 75 years of age.
2. aSAH patients with secured aneurysm.
3. Patient has cerebral vasospasm and is anesthetized and intubated.
4. Cerebral vasospasm is manifested by:

   * Mean Flow Velocity (MFV) >120 cm/sec in the intracranial ICA (Internal carotid artery), MCA (middle cerebral artery) or ACA (anterior cerebral artery) or MFV >110 cm/sec in the PCA, or >85 cm/sec in the vertebral or basilar arteries, as measured by TCD (Trans Cranial Doppler).

   Or:
   * Extra/intracranial ratio for the carotid watershed (MCA, ACA, intracranial ICA)>3, or a proximal/distal ratio for the vertebrobasilar (VB) system > 2.

   Or:
   * Affected/contralateral MCA MFV ratio ≥1.5. Or
   * Affected / baseline MCA MFV ratio ≥1.5.

   AND:
   * Vasoconstriction of at least 33% in at least one of the main cerebral arteries, measured by Angiography (Digital Subtraction Angiography (DSA) or Computed Tomography Angiography (CTA).
5. Hemodynamically stable, including subjects who are treated for fever, hydrocephalus, rebleeding, infection or metabolic abnormalities and are stable.
6. For pre-menopausal females - a negative pregnancy test, using an accepted method of birth control and avoid breast feeding for the duration of the trial
7. A legally Authorized representative have signed informed consent.

Exclusion Criteria:

1. WFNS score 5
2. Unsecured aneurysm or Intracranial/SAH of other than aneurysmal origin.
3. Signs attributable to serious aneurismal surgical procedure-related complications.
4. Patient underwent decompressive craniectomy.
5. S/p Carotid Endarterectomy, or other neck intervention.
6. Known carotid body tumor, past or present.
7. Hemodynamic instability due to cardiac arrhythmia or due to any other cause.
8. Had a myocardial infarction, unstable angina or syncope, congestive heart failure that require hospitalization or ejection fraction ≤ 40% within the past 3 months. Note: Elevated Troponin is expected after aSAH and will not exclude patients.
9. Had a stroke, within the past 1 year or transient ischemic attack at the last 3 months.
10. Any anatomical variation or thrombotic finding that according to the physician judgment is not eligible.
11. Renal insufficiency (Creatinine X2 of the normal).
12. Allergic to contrast media with no response to steroid pretreatment.
13. Are unable or unwilling to fulfill the protocol follow-up requirements
14. Are enrolled in another concurrent clinical trial, without prior approval of Samson NS and the PI.
15. Have an uncontrolled comorbid medical condition that would adversely affect their health if they are enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Device or procedure related (possibly, probably, or definitely) serious adverse events rate, from the treatment period and up to 30 days. | 30 days

SECONDARY OUTCOMES:
Decrease Mean Flow Velocity (MFV) of ≥15% below the maximal MVF measured prior to treatment, in at least one of the affected cerebral arteries, in at least one measuring during treatment | 7 days
Increase diameter of ≥15% in at least one of the affected main cerebral arteries, measured by Digital Subtraction Angiography (DSA) or Computed Tomography Angiography (CTA) | 7 days
Increase of ≥20% in PbtO2 above baseline prior to treatment measured by Licox® monitoring system during treatment | 7 days
Increase of ≥20% in CBF above baseline prior to treatment measured by the CerOx monitor system during treatment | 7 days
Mechanical performance of the Delta system | 7 days
  Lead shaft mechanical performance (e.g insertion, positioning/re positioning, fixation and retrieval) will be quantitatively measured
Electrical performance of the Delta system | 7 days
  Electrical performance of the electrical stimulation unit will be quantitatively measured

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vajkoczy, Prof., Principal Investigator — Charite - Universitätsmedizin, Department of Neurosurgery (Campus Virchow Klinikum), Berlin 113353, Germany
Locations (7):
- Czechia (2):
  - FN Brno, Jihlavská 20 625 00 Brno
  - UVN Praha Central Military Hospital, Prague
- Germany (4):
  - Charite Universitätsmedizin Berlin, Berlin
  - Johann Wolfgang Goethe-Universität, Frankfurt
  - Neurochirurgische Universitätsklinik Georg-August-Universität, Göttingen
  - University of Heidelberg, Heidelberg
- The Chaim Sheba Medical Center, Department of Neurosurgery, Tel Litwinsky, Israel